CLINICAL TRIAL: NCT03645967
Title: Efficacy of Meatal and Perineal Care With a Prepackaged Cleansing Cloth and Standardized Cleansing Protocol in Reducing Catheter-Associated Urinary Tract Infections in Acute-Care Hospitals
Brief Title: Efficacy of a Prepackaged Cleansing Cloth and Standardized Cleansing Protocol for Catheter Care at Reducing CAUTI Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R17-019
Record Dates: First submitted 2018-07-26; First posted 2018-08-24 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2021-10

CONDITIONS: Catheter-Associated Urinary Tract Infection

STUDY DESIGN:
Intervention Model Description: Intervention in the standard of care for indwelling urinary catheter care and maintenance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ReadyCleanse for IUC (Other): ReadyCleanse Cloths will be used for the standard of care for indwelling urinary catheter care and maintenance. The old standard of care will no longer be used.
  Interventions: Device: ReadyCleanse Cloths

INTERVENTIONS:
Device: ReadyCleanse Cloths — ReadyCleanse cloths and the standardized cleansing procedure will be the standard-of-care for catheter care and maintenance; patients will undergo routine perineal care for a minimum of twice per day and after each incontinent episode.

SUMMARY:
Superiority study evaluating the efficacy of a prepackaged cleansing cloth and standardizing cleansing protocol vs. previous standard-of-care for catheter care and maintenance.

DETAILED DESCRIPTION:
A superiority study evaluating the efficacy of a complete cleansing system composed of 5 prepackaged, moistened cloths with a standardized cleaning method compared to the previous standard-of-care for catheter care and maintenance. The primary objective is to investigate if the implementation of prepackaged cleansing cloths with a standardized cleaning protocol for all indwelling urinary catheter (IUC) care and maintenance provides a reduction in CAUTIs. The ReadyCleanse complete cleansing system will replace the previous standard-of-care. The ReadyCleanse intervention will be compared to the previous standard-of-care retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient who requires an IUC to be placed during admission to one of the four study hospitals

Exclusion Criteria:

* patients <18 years of age
* patients whose entire hospital stay occurs in: pediatric unit, psychiatric unit, labor & delivery or postpartum units, and emergency room

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9891 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal S Singh, MD, Principal Investigator — Endeavor Health
Locations (4):
- United States (4):
  - NorthShore University HealthSystem - Evanston, Evanston, Illinois
  - NorthShore University HealthSystem - Glenbrook, Glenview, Illinois
  - NorthShore University HealthSystem - Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem - Skokie, Skokie, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ReadyCleanse for IUC
Started | 9891
Completed | 9891
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ReadyCleanse for IUC
Number analyzed (Participants) | 9891
Age, Continuous [Mean (Full Range); unit: years] | 37.1 [24 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4540
  Male | 5351
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 457
  Native Hawaiian or Other Pacific Islander | 8
  Black or African American | 530
  White | 7105
  More than one race | 204
  Unknown or Not Reported | 1587
Region of Enrollment [Number; unit: participants]
  United States | 9891

OUTCOME MEASURES:

1. Primary Outcome: Infections Per 1,000 (CAUTI) Days
Description: Incidence Rate for CAUTIs per 1,000 Catheter days
Time Frame: 16 months
Measure: Number (95% Confidence Interval); unit: infection per 1,000 catheter days
Arm/Group | ReadyCleanse for IUC
Number analyzed (Participants) | 9872
infection per 1,000 catheter days | 0.8429 [0.6080 to 1.1685]

2. Secondary Outcome: Number of "Health Care Providers Responding to Health Care Provider Feedback Survey
Description: Healthcare provider feedback survey will be delivered to all staff that have utilized the ReadyCleanse cloths for indwelling urinary catheter care and maintenance. Purpose of the survey is to investigate healthcare provider preference and opinion of device.
Time Frame: Begins 3 months after start date. Time to take survey is approximately 10 minutes.
Population: Health Care Providers
Measure: Count of Participants; unit: Participants
Arm/Group | ReadyCleanse for IUC
Number analyzed (Participants) | 121
Participants | 121

ADVERSE EVENTS:
Time Frame: Participant Duration: Participant had an IUC inserted during their hospital stay, through study completion, an average of 4 days with 61 being the maximum number of days.
Description: If the condition of the participant's perineal skin and soft-tissue deteriorates unexpectedly, per the PI's interpretation, or if there is a new condition that the PI determines is not related to the baseline health condition but could be related to the use of the study product, it will be recorded as an AE.
Arm/Group | ReadyCleanse for IUC
All-Cause Mortality (participants affected / at risk) | 0/9872
Serious Adverse Events (participants affected / at risk) | 0/9872
Other Adverse Events (participants affected / at risk) | 0/9872

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03645967/Prot_SAP_000.pdf